CLINICAL TRIAL: NCT04255693
Title: Real-life Study of Changes of Gastroesophageal Reflux Disease Manifestations Due to Behavioural and Diet Adherence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Responsible Party: Principal Investigator, Sergey Morozov, Leading researcher, Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RLS-GERD
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Gastroesophageal Reflux Disease; GERD; Gastroesophageal Erosion; Erosive Esophagitis; Non-erosive Reflux Disease; Non-Erosive Gastro-Esophageal Reflux Disease
Keywords: GERD; NERD; erosive esophagitis; diet; food; adherence; influence
MeSH Terms: conditions — Gastroesophageal Reflux; Non-Erosive Reflux Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: According to the initial assessment, the patients will be allocated to the following subgroups: NERD, Erosive oesophagitis, hypersensitive oesophagus. Each patient will be provided with the standard recommendations on the diet and physical activity according to the initial assessment (calculated energy expenditures, physical activity, physical status and body composition) in addition to the standard drug treatment.
  Repeated examinations will be performed to assess the disease status and change (if any) of diet.
Who Masked: Outcomes Assessor
Masking Description: The personnel involved to the assessment of outcomes (changes in diet, changes on endoscopy, changes on symptoms) will be blinded to the results of each other.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Change in disease manifestations (Experimental): The data of all the patients will be assessed from the viewpoint of changes in the disease flow (severity and frequency of symptoms, grade of oesophagitis). They will be compared to the changes of the major factors that could influence the disease flow: adherence to anti-secretory agents, presence of concomitant medications and their doses, adherence to diet, change in physical activity. These will be compared to the initial data. Thus, it would be possible to make a multivariate comparison and try to establish the influence (and, possibly, weight) of each of the con-founder on the disease flow.
  Interventions: Behavioral: diet adherence; Behavioral: No diet adherence; Behavioral: Change in physical activity; Behavioral: No change in physical activity; Behavioral: Use of antisecretory agents; Behavioral: No use of antisecretory agents
- No change in disease flow (Active Comparator): To this arm patients with no change in the disease manifestations will be assigned, based on the end-point evaluation. The same as in the "experimental" groups factors will be analysed to establish the difference.
  Interventions: Behavioral: diet adherence; Behavioral: No diet adherence; Behavioral: Change in physical activity; Behavioral: No change in physical activity; Behavioral: Use of antisecretory agents; Behavioral: No use of antisecretory agents

INTERVENTIONS:
Behavioral: diet adherence — This type of "intervention" is to be established in a-posteriori analysis by the assessment of a fact whether a subject kept to use his "usual" diet or it contained substantial changes.
Behavioral: No diet adherence — A-posteriori established "intervention" based on the examinations at the end-point
Behavioral: Change in physical activity — The changes in physical activity will be assessed a-posteriori based on the examination at the end-point versus baseline data
Behavioral: No change in physical activity — The changes in physical activity will be assessed a-posteriori based on the examination at the end-point and comparison to the baseline data
Behavioral: Use of antisecretory agents — This "intervention" will be established a-posteriori, based on the examination at the end-point and compared to the baseline data. The need for the use of anti-secretory agents depends on the form of GERD and will be on the treating physician discretion. It is principal to account the use of anti-secretory agents (H2-histamine receptors blockers, proton pump inhibitors) as a major factors that may influence the outcomes.
Behavioral: No use of antisecretory agents — This "intervention" will be established a-posteriori, based on the examination at the end-point and compared to the baseline data.

SUMMARY:
This study is aimed to investigate the role of long-term diet adherence on manifestations of gastroesophageal reflux disease

DETAILED DESCRIPTION:
The role of diet in the treatment of gastroesophageal reflux disease (GERD) is still under discussion. Some studies support the evidence that specific components of food plays a role in triggering symptoms or may have an impact on reflux oesophagitis. Still, only limited data are present on the long-term real-life effects of diet and behaviour on the disease manifestations and outcomes. This specific study aims to investigate the role of diet in real-life cohort of patients in whom diagnosis of GERD is initially confirmed with the use of modern techniques (questionnaires, endoscopy, oesophageal pH-impedance recordings). To make the study possible, it is planned to form a cohort of patients with different manifestations of gastroesophageal reflux disease: non-erosive GERD (NERD), reflux-oesophagitis (EE), hypersensitive oesophagus. Each form of GERD is to be established in accordance to modern concept of GERD (i.e. Lyon consensus). In addition to standard-of-care examinations, diet assessment will be performed with the use of computer-based food frequency questionnaire (FFQ), which allows to analyse frequently used foods, food products in terms of frequency of consumption and sizes of the portions. Assessment of diet will be performed at the enrolment and than with a period of three months during three years. Based on the results, it would be possible to assess the effect of long-term adherence to diet, change of the composition of it, and perform a multifactorial statistical analysis with the consideration of other confounders: change in BMI, physical activity, smoking, concomitant medications, etc.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate (based on the signed informed consent form);
* presence of gastroesophageal reflux disease, based on the following: a) typical symptoms, like heartburn and/or regurgitation (for primary selection, symptoms should be present at least weekly, be actual for at least 3 months prior to the enrolment, and the patient should report the history of symptoms which lasts for at least 6 months); b) previous response to the intake of proton pump inhibitors; c) data of 24-hours oesophageal pH-impedance monitoring with detected pathological gastroesophageal reflux according to the Lyon consensus definitions;

Exclusion Criteria:

* pregnant or breast-feeding females;
* abdominal or chest surgery (except appendectomy or cholecystectomy in case they are not followed by adhesive disease of the abdominal organs);
* constant use of non-steroidal anti-inflammatory agents (NSAIDs), sporadic use of NSAIDs will be allowed in case the course of treatment was discontinued at least 2 weeks prior to the enrolment, in case that constant use of NSAIDs happen to be necessary after the enrolment, the patients may continue in the study but doses, frequency and duration of treatment should be carefully documented;
* history or current evidence of cancer of any aetiology and location besides skin cancer in situ successfully treated before the enrolment;
* severe patient's conditions which may lead to misinterpretation of data, or in case of patient's enrolment may put him at risk of exacerbation of co-morbid conditions, or in cases when on discretion of the investigator patient's condition would not allow him to complete the course of the observation. These conditions include, but not limited to: heart failure (class III-IV by NYHA), uncontrolled hypertension, severe neurological disorders, decompensated liver cirrhosis (Child-Pugh B or C), severe depression or other psychological disorders;
* the patient may stop his participation in the study at any time by informing the site personal about his/her decision to withdraw the consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Heartburn frequency | a week
  Number of days a week when the symptom is present
Heartburn severity | a day
  Subjective description reported by the patient, assessed with the use of visual analogue scale, from 0 to 5, where 0 is "not at all severe" and 5 is "very severe"
Grade of erosive oesophagitis | at the end-point, 2 years after enrolment
  Grade of oesophagitis will be assessed according to the Los-Angeles classification

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Morozov, MD, PhD, Principal Investigator — Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Locations (1):
- Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participants data may be shared by request. Patients personal data (name, contacts, etc) will be blinded beforehand, according to the law.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will be available when the study is accomplished. They will be available for the request for 2 years after the date of the study completion
Access Criteria: By request, when the reason for IPD sharing is reasonable and clear
URL: http://ion.ru

REFERENCES:
- [Background] Gyawali CP, Kahrilas PJ, Savarino E, Zerbib F, Mion F, Smout AJPM, Vaezi M, Sifrim D, Fox MR, Vela MF, Tutuian R, Tack J, Bredenoord AJ, Pandolfino J, Roman S. Modern diagnosis of GERD: the Lyon Consensus. Gut. 2018 Jul;67(7):1351-1362. doi: 10.1136/gutjnl-2017-314722. Epub 2018 Feb 3. PMID 29437910
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Savarino E, Bredenoord AJ, Fox M, Pandolfino JE, Roman S, Gyawali CP; International Working Group for Disorders of Gastrointestinal Motility and Function. Expert consensus document: Advances in the physiological assessment and diagnosis of GERD. Nat Rev Gastroenterol Hepatol. 2017 Nov;14(11):665-676. doi: 10.1038/nrgastro.2017.130. Epub 2017 Sep 27. PMID 28951582
- [Background] Roman S, Gyawali CP, Savarino E, Yadlapati R, Zerbib F, Wu J, Vela M, Tutuian R, Tatum R, Sifrim D, Keller J, Fox M, Pandolfino JE, Bredenoord AJ; GERD consensus group. Ambulatory reflux monitoring for diagnosis of gastro-esophageal reflux disease: Update of the Porto consensus and recommendations from an international consensus group. Neurogastroenterol Motil. 2017 Oct;29(10):1-15. doi: 10.1111/nmo.13067. Epub 2017 Mar 31. PMID 28370768
- [Background] Commisso A, Lim F. Lifestyle Modifications in Adults and Older Adults With Chronic Gastroesophageal Reflux Disease (GERD). Crit Care Nurs Q. 2019 Jan/Mar;42(1):64-74. doi: 10.1097/CNQ.0000000000000239. PMID 30507666
- [Background] Martinucci I, Natilli M, Lorenzoni V, Pappalardo L, Monreale A, Turchetti G, Pedreschi D, Marchi S, Barale R, de Bortoli N. Gastroesophageal reflux symptoms among Italian university students: epidemiology and dietary correlates using automatically recorded transactions. BMC Gastroenterol. 2018 Jul 17;18(1):116. doi: 10.1186/s12876-018-0832-9. PMID 30016938